CLINICAL TRIAL: NCT00588380
Title: A Pilot Study Examining How Common Genetic Variation in GLP1R Alters Response to GLP1 Infusion
Brief Title: GLP1R Polymorphisms and Response to GLP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Adrian Vella, Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07-004153
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Results first posted 2011-12-06 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Diabetes
Keywords: GLP-1; Insulin Secretion
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GLP-1 (Experimental): All participants recieved GLP-1 intravenously at 0.75 pmol/kg/min for the first hour and then at 1.5 pmol/kg/min for the next hour
  Interventions: Drug: GLP-1

INTERVENTIONS:
Drug: GLP-1 — GLP-1 infused at 0.75 pmol/kg/min from 121-180 minutes, GLP-1 infused at 1.55 pmol/kg/min from 181-240 minutes,

SUMMARY:
Glucagon-like Peptide-1 (GLP-1) is an important incretin hormone which acts as a powerful insulin secretagogue. Defects in GLP-1 synthesis and secretion are thought to be part of the pathogenesis of type 2 diabetes. Furthermore GLP-1 based therapy is an important part of the therapeutic armamentarium for the treatment of type 2 diabetes. The GLP-1 receptor (GLP1R) is the principal site of action of GLP-1 and GLP-1 receptor agonists like exenatide and liraglutide. The gene coding for this receptor, GLP1R, is highly polymorphic and contains numerous non-synonymous Single Nucleotide Polymorphisms (nsSNPs) which could potentially alter response to endogenous or exogenous GLP-1 or GLP-1R agonists. Indeed there is some in vitro data to support this concept. We propose to utilize a hyperglycemic clamp to test the insulin secretory response to infused GLP-1 in healthy volunteers to determine the effect of genetic variation in GLP1R on response to GLP-1.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40
* fasting glucose concentration of less than 95 mg/dl.

Exclusion Criteria:

* Individuals with a BMI < 19 or > 40 kg/m^2
* active systemic illness
* medication that can alter gastric emptying, insulin secretion & action
* history of abdominal surgery (other than appendectomy or tubal ligation).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Sathananthan A, Man CD, Micheletto F, Zinsmeister AR, Camilleri M, Giesler PD, Laugen JM, Toffolo G, Rizza RA, Cobelli C, Vella A. Common genetic variation in GLP1R and insulin secretion in response to exogenous GLP-1 in nondiabetic subjects: a pilot study. Diabetes Care. 2010 Sep;33(9):2074-6. doi: 10.2337/dc10-0200. PMID 20805279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers recruited from Olmsted County, MN.
Groups:
- Overall Study: All participants recieved glucose for 2 hours then Glucagon Like Peptide-1 (GLP-1) intravenously at a rate of 0.75 pmol/kg/min for 1 hour followed by 1.5 pmol/kg/min for the subsequent hour. The study lasted for 240 minutes.
Period: Overall Study
Arm/Group | Overall Study
Started | 88
Completed | 88
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 88
Age Continuous [Mean (Standard Deviation); unit: years] | 26.3 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 88

OUTCOME MEASURES:

1. Primary Outcome: Insulin Secretion at 150-180 Minutes.
Description: The 180 minute value represents the mean of the values obtained at 150, 160, 170, and 180 minutes.
Time Frame: 150 - 180 minutes after GLP-1 infusion
Population: all participants completed the study
Measure: Mean (Standard Error); unit: 10^-9 min^-1
Groups:
- All Participants: C-peptide as a marker of insulin secretion
Arm/Group | All Participants
Number analyzed (Participants) | 88
10^-9 min^-1
  rs6923761 (1,1) genotype | 104 (9)
  rs6923761 (1, 2) genotype | 94 (11)
  rs6923761 (2, 2) genotype | 81 (8)
  rs3765467 (1,2) genotype | 92 (6)
  rs3765467 (2,2) genotype | 219 (35)
Statistical Analysis 1: Comparison: All Participants; Using the Kruskal-Wallis test (general allelic model), we assessed univariate associations of rs6923761 genotype with Phi Total in the presence of either glucose alone, glucose and 0.75 pmol/kg/min GLP-1 or glucose and 1.5 pmol/kg/min GLP-1 If the p-value for the overall univariate test of association was <0.1, then the associations for specific genotype pairs (e.g.: 1,1 vs. 1,2 or 2,2 vs. 1,1) were also examined using a Mann-Whitney Rank Sum test; Test type: Superiority or Other; p = 0.11, Kruskal-Wallis

2. Secondary Outcome: Insulin Secretion at 210-240 Minutes
Description: The 240 minute value represents the mean of values obtained at 210, 220, 230, and 240 minutes.
Time Frame: 210 - 240 minutes after GLP-1 infusion
Population: All participants completing the study.
Measure: Mean (Standard Error); unit: 10^-9 min^-1
Arm/Group | Overall Study
Number analyzed (Participants) | 88
10^-9 min^-1
  rs6923761 (1,1) genotype | 152 (12)
  rs6923761 (1,2) genotype | 133 (15)
  rs6923761 (2,2) genotype | 112 (10)
  rs3765467 (1,2) genotype | 132 (7)
  rs3765467 (2,2) genotype | 325 (44)
Statistical Analysis 1: Comparison: Overall Study; All data are presented as means ± SEM. Using the Kruskal-Wallis test (general allelic model), we assessed univariate associations of genotype with ΦTotal; Test type: Superiority or Other; p = 0.09, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Duration of the study (4 hours)
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/88
Other Adverse Events (participants affected / at risk) | 0/88

LIMITATIONS AND CAVEATS:
This is a pilot study with limited power to detect / replicate effects. It will require independent replication of study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No